CLINICAL TRIAL: NCT01572493
Title: A Phase I Study of a Continuous Intravenous Infusion of Recombinant Human Interleukin IL-15 (rhIL-15) in Adults With Metastatic Cancers
Brief Title: Continuous Infusion of rhIL-15 for Adults With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kevin Conlon, MD, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 120113; 12-C-0113
Record Dates: First submitted 2012-04-05; First posted 2012-04-06 (Estimated); Results first posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Lymphoma; Carcinoma
Keywords: Pharmacokinetics of lL-15; Cytokine Therapy; Effects of rhlL-15 on T-cells and NK cells; Immunotherapy
MeSH Terms: conditions — Lymphoma; Carcinoma | interventions — Interleukin-15

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A1 (Dose Escalation, 10-day Dosing) (Experimental): Maximum tolerated dose (MTD) determination in subjects with metastatic cancers receiving recombinant human Interleukin-15 (rhIL-15) intravenous (IV) for 10 consecutive days
  Interventions: Biological: rh IL-15 (10 DAYS)
- Arm A2 (Dose Expansion, 10-day Dosing) (Experimental): Clinical activity evaluation in subjects with metastatic cancers receiving recombinant human Interleukin-15 (rhIL-15) intravenous (IV) for 10 consecutive days
  Interventions: Biological: rh IL-15 (5 DAYS)
- Arm B1 (Dose Escalation, 5-day Dosing) (Experimental): Maximum tolerated dose (MTD) determination in subjects with metastatic unresectable cancers receiving recombinant human Interleukin-15 (rhIL-15) intravenous (IV) for 5 consecutive days
  Interventions: Biological: rh IL-15 (5 DAYS)
- Arm B2 (Dose Expansion, 5-day Dosing) (Experimental): Clinical activity evaluation in subjects with metastatic cancers receiving recombinant human Interleukin-15 (rhIL-15) intravenous (IV) for 5 consecutive days
  Interventions: Biological: rh IL-15 (5 DAYS)

INTERVENTIONS:
Biological: rh IL-15 (10 DAYS) — Continuous infusion of recombinant human Interleukin-15 (rh IL-15) intravenous (IV) for first 10 days of each cycle
  Other Names: Recombinant human Interleukin-15
  Arms: Arm A1 (Dose Escalation, 10-day Dosing)
Biological: rh IL-15 (5 DAYS) — Continuous infusion of recombinant human Interleukin-15 (rh IL-15) for first 5 days of each cycle
  Other Names: Recombinant human Interleukin-15
  Arms: Arm A2 (Dose Expansion, 10-day Dosing); Arm B1 (Dose Escalation, 5-day Dosing); Arm B2 (Dose Expansion, 5-day Dosing)

SUMMARY:
Background:

- People with cancer can have a weak immune system as a result of the cancer itself, or from prior treatments. Still, treatments that stimulate the immune system have been shown to be effective against a number of different cancers. Recombinant human interleukin-15 (rhIL-15) is a drug that is designed to boost the immune system. Researchers are interested in seeing if rhIL-15 can strengthen the immune system's response against cancer. The drug will be given through a vein without a break for 10 days (240 hours).

Objectives:

* To see rhIL-15 given as a continuous infusion over 10 days can be used to treat advanced cancer
* Identify the side effects associated with this treatment.

Eligibility:

- Individuals at least 18 years of age with advanced cancer for which there are no effective treatments.

Design:

* Participants screening procedures will include a physical exam and medical history, laboratory (blood) tests and x-rays (Imaging studies) to determine suitability for the protocol.
* Appropriate participants with easily accessible tumor deposits may also be asked to have one pretreatment and one post (cycle 1) treatment tumor biopsy.
* Eligible participants will be admitted to the hospital for the rhIL-15 treatment and will spend about 12 days in the hospital.
* Participants will receive one 10 day infusion each cycle (about every 42 days) for as long as there are no serious side effects and the disease does not progress.
* Participants will continue treatment as long as imaging studies show that the tumor continues to shrink or for two additional cycles after it has disappeared from the x-rays to make that the cancer is completely gone.
* Participants who stop treatment for side effects or because their tumor did not shrink or stopped responding to the treatment will continue to have follow-up visits to monitor the outcome of the rhIL-15 treatment until there is evidence their cancer has progress or they begin another treatment.

DETAILED DESCRIPTION:
BACKGROUND:

* Interleukin-15 (IL-15) is a stimulatory cytokine with a number of desirable immunotherapeutic features, and clinical trials evaluating recombinant human interleukin-15 (rhIL-15) are underway.
* In contrast to IL-2, IL-15 treatment does not stimulate activation-induced cell death of T-cells; potentially inhibits immunosuppressive cluster of differentiation 4 (CD4) + Interleukin-2 receptor alpha chain (CD25) + T regulatory cells, contributes to the proliferation, differentiation and activation of CD8+ T-cells and NK-cells and the maintenance of long-term cluster of differentiation 8 (CD8) + memory T-cells.
* IL-15 is active in a number of syngeneic mouse preclinical tumor models, and vaccinia-based constructs expressing IL-15 induced long-lasting, high-avidity cytotoxic CD8+ T-lymphocyte response that appears to be more effective than similar IL-2 expressing vaccines.
* Pharmacology/toxicology (pharm/tox) experiments in non-human primate (NHP) rhesus macaques and preliminary results from the first-in-human phase I trial examining rhIL-15 given as an intravenous (IV) bolus (IVB) for 12 consecutive days indicate significant stimulation and expansion of NK-cells and CD8+ T-cells.
* rhIL-15 given as an IVB at 1 mcg/kg dose level appears to be well tolerated despite the presence of some common cytokine-related side effects indicating that 0.1 mcg/kg/day is an appropriate initial dose level for a phase I safety trial of continuous intravenous infusion (CIV) of rhIL-15.
* Comparison of the pharmacokinetic and immunologic assessments from the IVB phase I trial with the data from both sets of NHP pharm/tox experiments suggest that continuous intravenous (CIV) of rhIL-15 may have greater potential for stimulating an anticancer cellular immune response with a more manageable safety profile.

OBJECTIVES:

Primary Objective:

- Determine the safety, toxicity profile, dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) of rhIL-15 administered as a CIV for 10 consecutive days (240 hours) in subjects with metastatic unresectable cancers for which curative or palliative measures either do not exist or are not associated with a survival advantage.

ELIGIBILITY CRITERIA:

* Patients greater than or equal to18 years-old, Eastern Cooperative Oncology Group (ECOG) performance status (PS) less than or equal to 1, with pathologically confirmed metastatic unresectable cancers for which curative or palliative measures either do not exist or are not associated with a survival advantage.
* Patients with measurable or evaluable disease, normal organ and bone marrow function.

DESIGN:

* This is a single-institution, open-label, non-randomized 3 + 3 design phase I dose escalation study.
* Groups of 3 to 6 subjects will receive CIV rhIL-15 at doses of 0.1, 0.25, 0.5 1, 2, 4, 6 and 8 mcg/kg/day for 10 days provided that DLT has not been observed.
* After assessments of the 10-day dosing cohorts have been completed, new groups of 3 to 6 subjects will receive CIV rhIL-15 at doses of 3, 4 and 5 mcg/kg/day for 5 days provided that a DLT has not been observed.
* Patients with evidence of response and the absence of significant toxicities will be eligible for repeat cycles of treatment.
* Samples for correlative studies will be obtained prior to treatment and at specific times points during and after treatment to assess pharmacokinetics of rhIL-15, the effect of rhIL-15 on immune cell subset populations and pro-inflammatory cytokine levels in the peripheral blood and for the development of neutralizing anti-rhIL-15 antibodies.

ELIGIBILITY:
* INCLUSION CRITERIA
* Age greater than or equal to 18 years.
* Patients must have histologically confirmed (by the National Cancer Institute (NCI) Pathology Department) solid tumor malignancy or lymphoma that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are associated with minimal patient survival benefit (as defined the Metabolism Branch physicians or if the patient refuses standard of care treatment). Enrollment of patients with tumors that can be safely biopsied is encouraged.
* Patients must have evaluable or measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as greater than or equal to 20 mm with conventional techniques or as greater than or equal to 10 mm with spiral computed tomography (CT) scan.
* Patients must have recovered to < grade 1 Common Terminology Criteria for Adverse Events (CTCAE)v4 from toxicity of prior chemotherapy or biologic therapy and must not have had prior chemotherapy or biologic therapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C, 8 weeks for 7-hydroxystaurosporine (UCN-01).
* Patients must be at least 1 month since any prior radiation or major surgery.
* Patients on bisphosphonates for any cancer or on hormone therapy for prostate cancer will not need to discontinue this therapy to be eligible. However, patients with prostate cancer will need to have metastatic prostate cancer that has progressed despite hormonal therapy. Castrate testosterone levels occur within hours after castration and within 2 to 3 weeks of a luteinizing hormone-releasing hormone agonist. The current standard is to continue androgen suppression despite progressive disease.
* Diffusing capacity for carbon monoxide (DLCO)/alveolar volume (VA) and forced expiratory volume (FEV)-1.0 > 60% of predicted on pulmonary function tests.
* Serum creatinine of less than or equal to 1.5 X the upper limit of normal.
* Aspartate aminotransferase (AST) and alanine aminotransferase (AST) < 2.5 x the upper limit of normal.
* Absolute neutrophil count greater than or equal to 1,500/mm(3) and platelets greater than or equal to 100,000/mm(3).
* Karnofsky performance status greater than or equal to 70% or Eastern Cooperative Oncology Group (ECOG) less than or equal to 1
* Subjects with inactive central nervous system (CNS) metastasis are eligible. Inactive CNS metastasis is defined as: no signs of cerebral edema after successful definitive treatment of brain metastases (surgical resection, whole brain irradiation, stereotactic radiation therapy, or a combination of these) with stable or improved radiographic appearance on magnetic resonance imaging (MRI) scan at least 1 month after completion of treatment.

EXCLUSION CRITERIA:

* Patients who have received any systemic corticosteroid therapy within 3 weeks prior to the start of therapy with the exception of physiological replacement doses of cortisone acetate or equivalent.
* Patients who have received any cytotoxic therapy, immunotherapy, antitumor vaccines, monoclonal antibodies or major surgery in the 4 weeks prior to the start of the study.
* Life expectancy of less than 3 months.
* Patients with more than 30% replacement of hepatic parenchyma by tumor or any history of drug related hepatic encephalopathy.
* History of complex ventricular or supraventricular arrhythmias
* Documented human immunodeficiency virus (HIV), active bacterial infections, active or chronic hepatitis B, or hepatitis C infection.
* A positive hepatitis B serology indicative of previous immunization (i.e., hepatitis B surface antigen (HBsAb) positive and hepatitis B core antibody (HBcAb) negative), or a fully resolved acute hepatitis B infection is not an exclusion criterion.
* A positive hepatitis C serology is an exclusion criterion.
* Concurrent anticancer therapy (including other investigational agents), with the exception of hormone therapy for prostate cancer.
* Active central nervous system (CNS) metastases (inactive CNS metastases are defined).
* History of severe asthma or presently on chronic inhaled corticosteroid medications (patients with a history of mild asthma controlled with inhaled bronchodilators are eligible).
* History of autoimmune disease, with the exception of an autoimmune event associated with prior ipilimumab (anti-cluster of differentiation 152 (CTLA-4) therapy that has been completely resolved for more than 4 weeks.
* Inability or refusal to practice effective contraception during therapy or the presence of pregnancy or active breastfeeding (men and women of childbearing potential must use an effective method of birth control or abstinence during treatment and for 4 months after completion of treatment).
* Cognitive impairment, history of medical or psychiatric disease, other uncontrolled intercurrent illness, active substance abuse, or social circumstances, which in the view of the Principal Investigator (PI), would preclude safe treatment or the ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-04-04 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Conlon, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grabstein KH, Eisenman J, Shanebeck K, Rauch C, Srinivasan S, Fung V, Beers C, Richardson J, Schoenborn MA, Ahdieh M, et al. Cloning of a T cell growth factor that interacts with the beta chain of the interleukin-2 receptor. Science. 1994 May 13;264(5161):965-8. doi: 10.1126/science.8178155.
- [Background] Bamford RN, Grant AJ, Burton JD, Peters C, Kurys G, Goldman CK, Brennan J, Roessler E, Waldmann TA. The interleukin (IL) 2 receptor beta chain is shared by IL-2 and a cytokine, provisionally designated IL-T, that stimulates T-cell proliferation and the induction of lymphokine-activated killer cells. Proc Natl Acad Sci U S A. 1994 May 24;91(11):4940-4. doi: 10.1073/pnas.91.11.4940. PMID 8197161
- [Background] Burton JD, Bamford RN, Peters C, Grant AJ, Kurys G, Goldman CK, Brennan J, Roessler E, Waldmann TA. A lymphokine, provisionally designated interleukin T and produced by a human adult T-cell leukemia line, stimulates T-cell proliferation and the induction of lymphokine-activated killer cells. Proc Natl Acad Sci U S A. 1994 May 24;91(11):4935-9. doi: 10.1073/pnas.91.11.4935. PMID 8197160
- [Result] Conlon KC, Potter EL, Pittaluga S, Lee CR, Miljkovic MD, Fleisher TA, Dubois S, Bryant BR, Petrus M, Perera LP, Hsu J, Figg WD, Peer CJ, Shih JH, Yovandich JL, Creekmore SP, Roederer M, Waldmann TA. IL15 by Continuous Intravenous Infusion to Adult Patients with Solid Tumors in a Phase I Trial Induced Dramatic NK-Cell Subset Expansion. Clin Cancer Res. 2019 Aug 15;25(16):4945-4954. doi: 10.1158/1078-0432.CCR-18-3468. Epub 2019 May 29. PMID 31142503
- [Derived] Dubois SP, Miljkovic MD, Fleisher TA, Pittaluga S, Hsu-Albert J, Bryant BR, Petrus MN, Perera LP, Muller JR, Shih JH, Waldmann TA, Conlon KC. Short-course IL-15 given as a continuous infusion led to a massive expansion of effective NK cells: implications for combination therapy with antitumor antibodies. J Immunother Cancer. 2021 Apr;9(4):e002193. doi: 10.1136/jitc-2020-002193. PMID 33883258
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-C-0113.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were enrolled in the dose expansion phase of the study.
Groups:
- Dose Escalation Level 1 - 0.1 mcg/kg/Day x 10 Days: Level 1 - 0.1 mcg/kg/day x 10 Days
- Dose Escalation Level 2 - 0.25 mcg/kg/Day x 10 Days: Level 2 - 0.25 mcg/kg/day x 10 Days
- Dose Escalation Level 3 - 0.5 mcg/kg/Day x 10 Days: Level 3 - 0.5 mcg/kg/day x 10 Days
- Dose Escalation Level 4 - 1 mcg/kg/Day x 10 Days: Level 4 - 1 mcg/kg/day x 10 Days
- Dose Escalation Level 5 - 2 mcg/kg/Day x 10 Days: Level 5 - 2 mcg/kg/day x 10 Days
- Dose Escalation Level 6 - 4 mcg/kg/Day x 10 Days: Level 6 - 4 mcg/kg/day x 10 Days
- Dose Escalation Level 7 - 3 mcg/kg/Day x 5 Days: Level 7 - 3 mcg/kg/day x 5 Days
- Dose Escalation Level 8 - 4 mcg/kg/Day x 5 Days: Level 8 - 4 mcg/kg/day x 5 Days
- Dose Escalation Level 9 - 5 mcg/kg/Day x 5 Days: Level 9 - 5 mcg/kg/day x 5 Days
Period: Overall Study
Arm/Group | Dose Escalation Level 1 - 0.1 mcg/kg/Day x 10 Days | Dose Escalation Level 2 - 0.25 mcg/kg/Day x 10 Days | Dose Escalation Level 3 - 0.5 mcg/kg/Day x 10 Days | Dose Escalation Level 4 - 1 mcg/kg/Day x 10 Days | Dose Escalation Level 5 - 2 mcg/kg/Day x 10 Days | Dose Escalation Level 6 - 4 mcg/kg/Day x 10 Days | Dose Escalation Level 7 - 3 mcg/kg/Day x 5 Days | Dose Escalation Level 8 - 4 mcg/kg/Day x 5 Days | Dose Escalation Level 9 - 5 mcg/kg/Day x 5 Days
Started | 4 | 3 | 3 | 6 | 9 | 2 | 4 | 3 | 4
Completed | 3 | 2 | 1 | 4 | 7 | 1 | 1 | 3 | 2
Not Completed | 1 | 1 | 2 | 2 | 2 | 1 | 3 | 0 | 2
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Switched to alternative treatment | 0 | 1 | 2 | 1 | 2 | 0 | 2 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Level 1 - 0.1 mcg/kg/Day x 10 Days | Dose Escalation Level 2 - 0.25 mcg/kg/Day x 10 Days | Dose Escalation Level 3 - 0.5 mcg/kg/Day x 10 Days | Dose Escalation Level 4 - 1 mcg/kg/Day x 10 Days | Dose Escalation Level 5 - 2 mcg/kg/Day x 10 Days | Dose Escalation Level 6 - 4 mcg/kg/Day x 10 Days | Dose Escalation Level 7 - 3 mcg/kg/Day x 5 Days | Dose Escalation Level 8 - 4 mcg/kg/Day x 5 Days | Dose Escalation Level 9 - 5 mcg/kg/Day x 5 Days | Total
Number analyzed (Participants) | 4 | 3 | 3 | 6 | 9 | 2 | 4 | 3 | 4 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 1 | 6 | 4 | 2 | 2 | 2 | 3 | 24
  >=65 years | 3 | 0 | 2 | 0 | 5 | 0 | 2 | 1 | 1 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.63 (5.11) | 51.97 (7.26) | 55.83 (18.4) | 55.05 (5.82) | 56.58 (12.89) | 62.75 (2.33) | 60.05 (10.92) | 60.9 (5.42) | 61.15 (7.42) | 58.48 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 2 | 7 | 1 | 4 | 1 | 2 | 21
  Male | 3 | 2 | 1 | 4 | 2 | 1 | 0 | 2 | 2 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3 | 6 | 9 | 2 | 4 | 3 | 4 | 34
  Unknown or Not Reported | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 5
  White | 2 | 3 | 2 | 4 | 6 | 2 | 4 | 2 | 4 | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 3 | 6 | 9 | 2 | 4 | 3 | 4 | 38
Diagnosis [Count of Participants; unit: Participants]
  Head and Neck cancer | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3
  Sarcoma | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 4
  Renal Cell carcinoma | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 4
  Pancreatic cancer | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 3
  Colorectal cancer | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 7
  Metastatic Melanoma | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
  Non-Small Cell Lung cancer (NSCLC) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
  Endometrial | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Adrenal | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Adenoid Cystic | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cholangiocarcinoma | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Gastric neuro-ectodermal | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Prostate | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
  Gastrointestinal Stromal Tumor | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Small bowel | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Esophageal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Performance Status - Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants] — Performance status ECOG 0 is normal activity, and 1 is symptoms, but ambulatory.
  Participants
    0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    1 | 4 | 3 | 3 | 6 | 9 | 2 | 4 | 3 | 4 | 38
Prior Therapy [Count of Participants; unit: Participants]
  Surgery | 3 | 2 | 2 | 5 | 3 | 2 | 4 | 2 | 3 | 26
  Chemotherapy | 3 | 3 | 1 | 5 | 4 | 2 | 4 | 3 | 3 | 28
  Radiation Therapy | 3 | 3 | 2 | 3 | 3 | 1 | 1 | 1 | 1 | 18
  Molecular Therapy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Immunotherapy | 2 | 2 | 0 | 1 | 3 | 1 | 1 | 3 | 1 | 14
  Checkpoint Inhibitors | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hormonal Therapy | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Recombinant Human Interleukin-15 (rhIL-15) for 10 Day Dosing
Description: The MTD is the dose level at which less than one-third of patients (0/3 or 0-1/6 participants) treated at that dose experience a dose-limiting toxicity (DLT), with the next higher dose level demonstrating a one-third or greater number of participants (≥ 2/3 or ≥ 2/6 participants) having DLT. A DLT is Grade 2 diarrhea lasting more than 24 hours or any grade 3 or 4 toxicity, if deemed possibly, probably or definitely related to the study drug by the principal investigator during the first cycle of treatment. Toxicities were assessed by the Common Terminology Criteria for Adverse Events (CTCAE)v4. Grade 3 is severe, and Grade 4 is life-threatening.
Time Frame: After one cycle (one cycle is 42 days for 10-day dosing)
Measure: Number; unit: mcg/kg/day
Groups:
- All Participants: All participants on the following dose levels:
  Level 1 - 0.1 mcg/kg/day x 10 Days Level 2 - 0.25 mcg/kg/day x 10 Days Level 3 - 0.5 mcg/kg/day x 10 Days Level 4 - 1 mcg/kg/day x 10 Days Level 5 - 2 mcg/kg/day x 10 Days Level 6 - 4 mcg/kg/day x 10 Days
Arm/Group | All Participants
Number analyzed (Participants) | 27
mcg/kg/day | 2

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Recombinant Human Interleukin-15 (rhIL-15) for 5 Day Dosing
Description: as for outcome 1
Time Frame: After one cycle (one cycle is 21 days for 5-day dosing)
Measure: Number; unit: mcg/kg/day
Groups:
- All Participants: All participants on the following dose levels:
  Level 7 - 3 mcg/kg/day x 5 Days Level 8 - 4 mcg/kg/day x 5 Days Level 9 - 5 mcg/kg/day x 5 Days
Arm/Group | All Participants
Number analyzed (Participants) | 9
mcg/kg/day | NA — The protocol stated that only if there was a clinical response in the 5-day cohorts, would a dose expansion cohort (and additional higher doses) be attempted. By this time about 70 participants had received the NCI rhIL-15 and there were no clinical responses and participants at the 4 and 5 mcg/kg/day were starting to demonstrate (non-DLT) pulmonary toxicity. So we had the information we needed for the "RPh2 dose."

3. Primary Outcome: Number of Participants With Grades 3, 4 or 5 Dose-Limiting Toxicity (DLT) Related to Study Drug
Description: A DLT is Grade 2 diarrhea lasting more than 24 hours or any grade 3 or 4 toxicity, if deemed possibly, probable or definitely related to the study drug by the principal investigator during the first cycle of treatment; and/or Grade 5 death related to adverse event. Toxicities were assessed by the Common Terminology Criteria for Adverse Events (CTCAE)v4. Grade 3 is severe, and Grade 4 is life-threatening.
Time Frame: After one cycle (one cycle is either 42 or 21 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Level 1 - 0.1 mcg/kg/Day x 10 Days | Dose Escalation Level 2 - 0.25 mcg/kg/Day x 10 Days | Dose Escalation Level 3 - 0.5 mcg/kg/Day x 10 Days | Dose Escalation Level 4 - 1 mcg/kg/Day x 10 Days | Dose Escalation Level 5 - 2 mcg/kg/Day x 10 Days | Dose Escalation Level 6 - 4 mcg/kg/Day x 10 Days | Dose Escalation Level 7 - 3 mcg/kg/Day x 5 Days | Dose Escalation Level 8 - 4 mcg/kg/Day x 5 Days | Dose Escalation Level 9 - 5 mcg/kg/Day x 5 Days
Number analyzed (Participants) | 4 | 3 | 3 | 6 | 9 | 2 | 4 | 3 | 4
Participants
  Grade 3 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

4. Secondary Outcome: Clinical Response Rate
Description: Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Complete response (CR) is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Progressive disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study, and the appearance of one or more new lesions. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Both cycles 1 and 2 (each cycle is 42 days) for the 10 day treatment, up to 84 days. And clinical responses for the 5-day treatment cohorts (21 day cycle length) were assessed after cycles 2, 4, 6, 8 and so on treatment cycles.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Level 1 - 0.1 mcg/kg/Day x 10 Days | Dose Escalation Level 2 - 0.25 mcg/kg/Day x 10 Days | Dose Escalation Level 3 - 0.5 mcg/kg/Day x 10 Days | Dose Escalation Level 4 - 1 mcg/kg/Day x 10 Days | Dose Escalation Level 5 - 2 mcg/kg/Day x 10 Days | Dose Escalation Level 6 - 4 mcg/kg/Day x 10 Days | Dose Escalation Level 7 - 3 mcg/kg/Day x 5 Days | Dose Escalation Level 8 - 4 mcg/kg/Day x 5 Days | Dose Escalation Level 9 - 5 mcg/kg/Day x 5 Days
Number analyzed (Participants) | 4 | 3 | 3 | 6 | 9 | 2 | 4 | 3 | 4
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Progressive Disease | 1 | 3 | 1 | 2 | 3 | 2 | 1 | 2 | 3
  Stable Disease | 2 | 0 | 2 | 3 | 4 | 0 | 2 | 1 | 0
  Not Assessed | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1

5. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the date of protocol consent until date of progressive disease is documented. Progressive disease was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Progressive disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study, and the appearance of one or more new lesions.
Time Frame: From the date of protocol consent until date of progressive disease is documented, up to 263 days
Population: One participant in dose level 1 and dose level 2, two participants in dose level 3, three participants in dose level 4, two participants in dose level 5, one participant in dose level 6 and dose level 7, and one participant in dose level 9 were not evaluable.
Measure: Median (Full Range); unit: Days
Groups:
- Dose Escalation Dose Escalation Level 7 - 3 mcg/kg/Day x 5 Days: Level 7 - 3 mcg/kg/day x 5 Days
Arm/Group | Dose Escalation Level 1 - 0.1 mcg/kg/Day x 10 Days | Dose Escalation Level 2 - 0.25 mcg/kg/Day x 10 Days | Dose Escalation Level 3 - 0.5 mcg/kg/Day x 10 Days | Dose Escalation Level 4 - 1 mcg/kg/Day x 10 Days | Dose Escalation Level 5 - 2 mcg/kg/Day x 10 Days | Dose Escalation Level 6 - 4 mcg/kg/Day x 10 Days | Dose Escalation Dose Escalation Level 7 - 3 mcg/kg/Day x 5 Days | Dose Escalation Level 8 - 4 mcg/kg/Day x 5 Days | Dose Escalation Level 9 - 5 mcg/kg/Day x 5 Days
Number analyzed (Participants) | 3 | 2 | 1 | 3 | 7 | 1 | 3 | 3 | 3
Days | 74 [28 to 138] | 54 [37 to 71] | 29 [NA to NA] — Data is for a single participant. | 77 [70 to 263] | 68 [30 to 74] | 6 [NA to NA] — Data is for a single participant. | 87 [49 to 91] | 42 [42 to 74] | 34.5 [9 to 42]

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Recombinant Human Interleukin-15 (rhIL-15)
Description: The maximum observed analyte concentration in serum was reported.
Time Frame: Prior to 1st dose, at 10 minutes after 1st dose, once daily on days 7-10 at completion of treatment, at 10 and 30 minutes after completion of treatment and at 1, 2, 4, and approximately 24 hours after completion of treatment.
Population: 3/4 participants in dose level 1, and 2/3 participants in dose level 2 were not evaluable for this outcome measure. Cmax was only performed for the 10 day dosing cohorts.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Dose Escalation Level 1 - 0.1 mcg/kg/Day x 10 Days | Dose Escalation Level 2 - 0.25 mcg/kg/Day x 10 Days | Dose Escalation Level 3 - 0.5 mcg/kg/Day x 10 Days | Dose Escalation Level 4 - 1 mcg/kg/Day x 10 Days | Dose Escalation Level 5 - 2 mcg/kg/Day x 10 Days | Dose Escalation Level 6 - 4 mcg/kg/Day x 10 Days
Number analyzed (Participants) | 1 | 1 | 3 | 6 | 9 | 2
pg/mL | 51 (NA) — Cannot determine geometric coefficient of variation value with one participant. | 59 (NA) — Cannot determine geometric coefficient of variation value with one participant. | 116 (72) | 1413 (1478) | 5662 (5961) | 26852 (11374)

7. Secondary Outcome: Concentration of Drug in Plasma at Steady State (Css)
Description: Concentration of drug in plasma at steady state (Css).
Time Frame: Days 7 through 10
Population: 3/4 participants in dose level 1, and 2/3 participants in dose level 2 were not evaluable for this outcome measure. Css was only performed for the 10 day dosing cohorts.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Dose Escalation Level 1 - 0.1 mcg/kg/Day x 10 Days | Dose Escalation Level 2 - 0.25 mcg/kg/Day x 10 Days | Dose Escalation Level 3 - 0.5 mcg/kg/Day x 10 Days | Dose Escalation Level 4 - 1 mcg/kg/Day x 10 Days | Dose Escalation Level 5 - 2 mcg/kg/Day x 10 Days | Dose Escalation Level 6 - 4 mcg/kg/Day x 10 Days
Number analyzed (Participants) | 1 | 1 | 3 | 6 | 9 | 2
pg/mL | 44.5 (NA) — Cannot determine geometric coefficient of variation value with one participant. | 48.5 (NA) — Cannot determine geometric coefficient of variation value with one participant. | 73.2 (22.6) | 489 (463) | 2020 (2309) | 9562 (59.35)

8. Secondary Outcome: Area Under the Curve (AUClast)
Description: AUClast is from dosing to the time of the last measured concentration >/= lower limit of quantitation (LLOQ)(Clast) of that dosing period.
Time Frame: as for outcome 6
Population: 3/4 participants in dose level 1, and 2/3 participants in dose level 2 were not evaluable for this outcome measure. AUClast was only performed for the 10 day dosing cohorts.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Dose Escalation Level 1 - 0.1 mcg/kg/Day x 10 Days | Dose Escalation Level 2 - 0.25 mcg/kg/Day x 10 Days | Dose Escalation Level 3 - 0.5 mcg/kg/Day x 10 Days | Dose Escalation Level 4 - 1 mcg/kg/Day x 10 Days | Dose Escalation Level 5 - 2 mcg/kg/Day x 10 Days | Dose Escalation Level 6 - 4 mcg/kg/Day x 10 Days
Number analyzed (Participants) | 1 | 1 | 3 | 6 | 9 | 2
pg/mL | 7756 (NA) — Cannot determine geometric coefficient of variation value with one participant. | 10907 (NA) — Cannot determine geometric coefficient of variation value with one participant. | 20798 (8667) | 187453 (206143) | 321747 (300686) | 262651 (77613)

9. Secondary Outcome: Inflammatory Cytokines
Description: Serum samples was obtained from participants and inflammatory cytokine analyses was performed by flow cytometry to determine levels of Interleukin - 1, Interferon γ, Interleukin-6 and Tumor Necrosis Factor ἁ.
Time Frame: Pre, 0.16, 1, 2, 4, 8, 12, and 24 hours on Day 1. Days 2, 7, 8, 9, and 10. 0, 0.16, 0.32, 1, 2, 4, and 12 hours on Day 11. And 24 hours on Day 12.
Population: This outcome measure was only performed for 10 day dosing.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Dose Escalation Level 1 - 0.1 mcg/kg/Day x 10 Days | Dose Escalation Level 2 - 0.25 mcg/kg/Day x 10 Days | Dose Escalation Level 3 - 0.5 mcg/kg/Day x 10 Days | Dose Escalation Level 4 - 1 mcg/kg/Day x 10 Days | Dose Escalation Level 5 - 2 mcg/kg/Day x 10 Days | Dose Escalation Level 6 - 4 mcg/kg/Day x 10 Days
Number analyzed (Participants) | 4 | 3 | 3 | 6 | 9 | 2
pg/mL
  Interleukin - 1, Pre Day 1 | 0.38 (0.24) | 0.24 (0) | 9.8 (15.9) | 0.86 (0.8) | 0.34 (0.1) | 0.24 (0)
  Interleukin - 1, 0.16 hours on Day 1 | 0.28 (0) | 0.24 (0) | 2.2 (3) | 19 (45) | 77 (229) | 0.24 (0)
  Interleukin - 1, 1 hour on Day 1 | 0.47 (0.3) | 0.24 (0) | 17.9 (30) | 9.1 (20) | 57 (170) | 0.24 (0)
  Interleukin - 1, 2 hours on Day 1 | 0.58 (0.3) | 0.24 (0) | 4.4 (6.8) | 3.5 (8) | 22 (65) | 0.24 (0)
  Interleukin - 1, 4 hours on Day 1 | 0.59 (0.3) | 0.24 (0) | 13.4 (21) | 0.53 (0.3) | 6.3 (16) | 0.36 (0.2)
  Interleukin - 1, 8 hours on Day 1 | 0.73 (0.1) | 0.24 (0) | 1.3 (1.4) | 0.83 (0.8) | 209 (605) | 0.24 (0)
  Interleukin - 1, 12 hours on Day 1 | 0.54 (0.2) | 0.24 (0) | 0.36 (0.2) | 0.5 (0.3) | 7 (19.7) | 0.24 (0)
  Interleukin - 1, 24 hours on Day 1 | 0.36 (0.2) | 0.24 (0) | 0.62 (0.65) | 1.2 (1.4) | 4.3 (8) | 0.24 (0)
  Interleukin - 1 on Day 2 | 0.42 (0.3) | 0.24 (0) | 0.94 (1.2) | 0.43 (0.3) | 1.1 (1.5) | 0.7 (0.6)
  Interleukin - 1 on Day 7 | 1.18 (0.9) | 0.24 (0) | 0.44 (0.35) | 0.32 (0.1) | 0.27 (0.1) | NA (NA) — tests not performed
  Interleukin - 1 on Day 8 | 0.43 (0.3) | 0.24 (0) | 0.25 (0.2) | 0.36 (0.3) | 0.29 (0.1) | NA (NA) — tests not performed
  Interleukin - 1 on Day 9 | 0.54 (0.5) | 0.24 (0) | 0.76 (0.23) | 0.38 (0.3) | 0.42 (0.4) | NA (NA) — tests not performed
  Interleukin - 1 on Day 10 | 0.45 (0.3) | 0.24 (0) | 0.59 (0.13) | 0.3 (0.1) | 0.37 (0.2) | NA (NA) — tests not performed
  Interleukin - 1, 0 hours on Day 11 | 0.72 (0.8) | 0.27 (0) | 0.69 (0.21) | 1.1 (0.8) | 0.62 (0.6) | NA (NA) — tests not performed
  Interleukin - 1, 0.16 hours on Day 11 | 0.62 (0.6) | 2.98 (4.7) | 0.64 (0.21) | 0.72 (0.4) | 0.61 (0.6) | NA (NA) — tests not performed
  Interleukin - 1, 0.32 hours on Day 11 | 0.69 (0.7) | 0.26 (0.4) | 0.56 (0.16) | 0.65 (0.5) | 0.56 (0.4) | NA (NA) — tests not performed
  Interleukin - 1, 1 hour on Day 11 | 8.69 (13.3) | 0.81 (0.9) | 0.45 (0.1) | 0.75 (0.6) | 0.6 (0.5) | NA (NA) — tests not performed
  Interleukin - 1, 2 hours on Day 11 | 0.51 (0.3) | 0.24 (0) | NA (NA) — tests not performed | 2.17 (1.7) | 0.52 (0.4) | NA (NA) — tests not performed
  Interleukin - 1, 4 hours on Day 11 | 1.2 (1.1) | 0.32 (0.1) | 16.2 (0) | 0.75 (0.6) | 0.42 (0.3) | NA (NA) — tests not performed
  Interleukin - 1, 12 hours on Day 11 | NA (NA) — tests not performed | 0.81 (0.6) | NA (NA) — tests not performed | NA (NA) — tests not performed | NA (NA) — tests not performed | NA (NA) — tests not performed
  Interleukin - 1, 24 hours on Day 12 | 0.44 (0.3) | 0.24 (0) | 16.2 (27) | 0.34 (0.1) | 0.27 (0.1) | NA (NA) — tests not performed
  Interferon γ, Pre Day 1 | 6.8 (6.9) | 4.6 (1.6) | 8.3 (8.9) | 4.7 (3) | 9.2 (6.3) | 2.8 (1)
  Interferon γ - 0.16 hours on Day 1 | 2.5 (1.6) | 3.4 (0.5) | 5.7 (4.7) | 17 (23) | 21 (40) | 1.72 (0)
  Interferon γ - 1 hour on Day 1 | 6.5 (5.5) | 4 (1) | 8.4 (8) | 4 (3.3) | 10.6 (10) | 2.9 (1.9)
  Interferon γ - 2 hours on Day 1 | 6.8 (5.9) | 4.7 (1.6) | 6.9 (4.4) | 4.5 (2.9) | 11.5 (7.2) | 7 (2)
  Interferon γ - 4 hours on Day 1 | 9.4 (6.8) | 4.9 (1) | 6.8 (3.2) | 11 (7) | 131 (289) | 131 (3.3)
  Interferon γ - 8 hours on Day 1 | 27 (14) | 5 (2.2) | 10.6 (6.5) | 24 (20) | 110 (170) | 97 (67)
  Interferon γ - 12 hours on Day 1 | 22.7 (24) | 5.7 (2) | 11.2 (7.4) | 29 (14.7) | 66.6 (39) | 38.7 (13)
  Interferon γ - 24 hours on Day 1 | 24.6 (34) | 6.6 (1.1) | 13.3 (8) | 32.8 (19) | 106 (84) | 94.6 (38)
  Interferon γ on Day 2 | 11.1 (12) | 8.1 (2.3) | 17 (10.1) | 58.4 (47) | 230 (205) | 639 (678)
  Interferon γ on Day 7 | 10 (10) | 8.6 (1.3) | 56 (55) | 43.8 (29) | 136 (74) | NA (NA) — tests not performed
  Interferon γ on Day 8 | 13.2 (18) | 9.5 (0.4) | 55.7 (57) | 52.9 (36) | 145 (109) | NA (NA) — tests not performed
  Interferon γ on Day 9 | 15 (20) | 8.9 (2.3) | 26.8 (21) | 132 (183) | 149 (112) | NA (NA) — tests not performed
  Interferon γ on Day 10 | 13.3 (16) | 8.9 (1.9) | 43 (10.7) | 262 (432) | 238 (214) | NA (NA) — tests not performed
  Interferon γ - 0 hours on Day 11 | 11 (11.4) | 7.8 (1) | 57.4 (34) | 451 (794) | 315 (327) | NA (NA) — tests not performed
  Interferon γ - 0.16 hours on Day 11 | 11.3 (12) | 7.7 (0.3) | 37.8 (6) | 99 (111) | 223 (180) | NA (NA) — tests not performed
  Interferon γ - 0.32 hours on Day 11 | 11.6 (12) | 7.6 (0.5) | 41 (1.1) | 101 (123) | 207 (177) | NA (NA) — tests not performed
  Interferon γ - 1 hour on Day 11 | 12 (12.4) | 7.5 (0.3) | 37.5 (4.7) | 106 (119) | 204 (172) | NA (NA) — tests not performed
  Interferon γ - 2 hours on Day 11 | 8.6 (8) | 5.5 (0.5) | 25.3 (0.5) | 96.6 (93) | 101 (170) | NA (NA) — tests not performed
  Interferon γ - 4 hours on Day 11 | 12.5 (13) | 7.6 (1.3) | 36.9 (10) | 89 (77) | 190 (141) | NA (NA) — tests not performed
  Interferon γ - 12 hours on Day 11 | NA (NA) — tests not performed | NA (NA) — tests not performed | NA (NA) — tests not performed | NA (NA) — tests not performed | NA (NA) — tests not performed | NA (NA) — tests not performed
  Interferon γ - 24 hours on Day 12 | 8.3 (84.6) | 5.1 (0.2) | 19 (6.4) | 27.4 (27) | 97 (145) | NA (NA) — tests not performed
  Interleukin-6, Pre Day 1 | 3.4 (2.6) | 5.3 (4.2) | 200 (342) | 2.1 (1.2) | 7.1 (9.6) | 4.6 (4.7)
  Interleukin-6 - 0.16 hours on Day 1 | 3.4 (2.4) | 5.3 (3.7) | 348 (596) | 6.2 (6.4) | 232 (682) | 6.8 (0)
  Interleukin-6 - 1 hour on Day 1 | 3.7 (3.8) | 5.2 (4.2) | 179 (303) | 3.7 (3.7) | 262 (773) | 3.9 (3.7)
  Interleukin-6 - 2 hours on Day 1 | 4.1 (4.2) | 6.6 (5.4) | 18.1 (23) | 3.2 (2.2) | 120 (349) | 3.8 (3.5)
  Interleukin-6 - 4 hours on Day 1 | 5.1 (4.3) | 6.9 (5.8) | 78 (127) | 2.9 (1.6) | 23.7 (30) | 45.6 (59)
  Interleukin-6 - 8 hours on Day 1 | 3 (0.45) | 6.6 (5.4) | 4.9 (2.5) | 6.6 (3.4) | 607 (1767) | 16.9 (9.4)
  Interleukin-6 - 12 hours on Day 1 | 6.3 (7) | 6.7 (5.9) | 4.4 (1.1) | 5.1 (3) | 18.4 (27) | 7.3 (4.8)
  Interleukin-6 - 24 hours on Day 1 | 4 (2.3) | 7.2 (5.8) | 5.1 (3.2) | 4.7 (1.9) | 19 (24) | 12.7 (10)
  Interleukin-6 on Day 2 | 2.2 (0.7) | 6.2 (4.5) | 6.2 (5.3) | 3.4 (1.7) | 13.2 (14) | 141 (112)
  Interleukin-6 on Day 7 | 15.2 (17) | 4.8 (2.8) | 6.6 (4.9) | 3.2 (0.9) | 8 (7.2) | NA (NA) — tests not performed
  Interleukin-6 on Day 8 | 4 (4.4) | 6.1 (4.1) | 2.9 (1.2) | 4.3 (1.9) | 8.8 (9.1) | NA (NA) — tests not performed
  Interleukin-6 on Day 9 | 3.4 (2.5) | 6.8 (5.4) | 5.2 (5.2) | 4.7 (2) | 9.9 (9.2) | NA (NA) — tests not performed
  Interleukin-6 on Day 10 | 3.8 (2.4) | 5.9 (4.7) | 3.1 (1) | 5.6 (3.1) | 12 (14) | NA (NA) — tests not performed
  Interleukin-6 - 0 hours on Day 11 | 3.7 (2.4) | 7.7 (6.3) | 11.6 (12) | 7.1 (7.6) | 10.2 (8.6) | NA (NA) — tests not performed
  Interleukin-6 - 0.16 hours on Day 11 | 3.6 (1.5) | 6.8 (6.2) | 16.3 (12.) | 7.9 (8.9) | 11.4 (9.7) | NA (NA) — tests not performed
  Interleukin-6 - 0.32 hours on Day 11 | 3.4 (1.4) | 113 (184) | 19.7 (13) | 5.1 (1.8) | 11.4 (9.2) | NA (NA) — tests not performed
  Interleukin-6 - 1 hour on Day 11 | 82 (136) | 6.8 (6.2) | 16 (13.5) | 5.1 (1.8) | 11.2 (8.9) | NA (NA) — tests not performed
  Interleukin-6 - 2 hours on Day 11 | 5.5 (4) | 45.7 (66) | 14.6 (10.) | 12.2 (16) | 11.4 (10) | NA (NA) — tests not performed
  Interleukin-6 - 4 hours on Day 11 | 3.7 (1.3) | 8.5 (7.6) | 13.3 (10) | NA (NA) — tests not performed | 9.8 (8.8) | NA (NA) — tests not performed
  Interleukin-6 - 12 hours on Day 11 | NA (NA) — tests not performed | NA (NA) — tests not performed | NA (NA) — tests not performed | NA (NA) — tests not performed | NA (NA) — tests not performed | NA (NA) — tests not performed
  Interleukin-6 - 24 hours on Day 12 | 2.9 (0.7) | 7.7 (6.6) | 30.4 (27) | 3.3 (1.1) | 8.3 (9.38) | NA (NA) — tests not performed
  Tumor Necrosis Factor ἁ, Pre Day 1 | 1.85 (0.8) | 2.3 (0.5) | 12.4 (18) | 2.2 (0.9) | 2.4 (0.6) | 1.8 (0.5)
  Tumor Necrosis Factor ἁ - 0.16 hours on Day 1 | 1.2 (0.4) | 1.7 (0.7) | 39 (66) | 3.40 (2) | 13.5 (34) | 1.9 (0)
  Tumor Necrosis Factor ἁ - 1 hour on Day 1 | 1.7 (0.8) | 2.3 (1.2) | 24 (39) | 2.7 (1.7) | 11.2 (27) | 1.7 (0.4)
  Tumor Necrosis Factor ἁ - 2 hours on Day 1 | 1.8 (1.0) | 2.4 (1.4) | 6.3 (8) | 2.5 (1) | 7.8 (15) | 2.5 (0.6)
  Tumor Necrosis Factor ἁ - 4 hours on Day 1 | 2.7 (1.7) | 2.2 (1.1) | 16 (25) | 2.9 (1.2) | 5.5 (3.7) | 6 (1.2)
  Tumor Necrosis Factor ἁ - 8 hours on Day 1 | 1.7 (0.5) | 2.4 (1.3) | 3.6 (2.2) | 4.3 (1.7) | 13.3 (20) | 6 (3)
  Tumor Necrosis Factor ἁ - 12 hours on Day 1 | 2.5 (1) | 2.6 (1.2) | 3.9 (2.4) | 5 (1.9) | 8.6 (3.3) | 6.3 (0.5)
  Tumor Necrosis Factor ἁ - 24 hours on Day 1 | 2.1 (0.5) | 2.9 (0.7) | 4.4 (3.3) | 6.4 (2.1) | 11.5 (6.4) | 9.2 (2.8)
  Tumor Necrosis Factor ἁ Day 2 | 2.3 (0.7) | 3.6 (0.4) | 5.1 (2.8) | 6.8 (2.3) | 11.6 (4.7) | 24 (7)
  Tumor Necrosis Factor ἁ on Day 7 | 2.9 (0.5) | 3 (1.2) | 5.5 (4.5) | 7.5 (2.1) | 13.8 (2.7) | NA (NA) — tests not performed
  Tumor Necrosis Factor ἁ on Day 8 | 2.7 (0.9) | 3.5 (1.5) | 5.6 (4.3) | 7.7 (2) | 13.4 (2.9) | NA (NA) — tests not performed
  Tumor Necrosis Factor ἁ on Day 9 | 2.6 (1.2) | 3.4 (1.6) | 5.3 (3.3) | 6.6 (2.7) | 11.2 (3.7) | NA (NA) — tests not performed
  Tumor Necrosis Factor ἁ on Day 10 | 2.7 (1.6) | 2.8 (1.4) | 5.6 (3.8) | 7.4 (2) | 11.1 (3.6) | NA (NA) — tests not performed
  Tumor Necrosis Factor ἁ - 0 hours on Day 11 | 2.4 (1.2) | 2.9 (1) | 6.3 (1.9) | 6.6 (1.7) | 10.7 (3) | NA (NA) — tests not performed
  Tumor Necrosis Factor ἁ - 0.16 hours on Day 11 | 2.2 (0.6) | 3 (1.2) | 4.7 (1.6) | 6.5 (1.6) | 9.8 (2.4) | NA (NA) — tests not performed
  Tumor Necrosis Factor ἁ - 0.32 hours on Day 11 | 2.5 (1.5) | 14.2 (20) | 5.5 (2.9) | 6 (1.3) | 9.4 (2.3) | NA (NA) — tests not performed
  Tumor Necrosis Factor ἁ - 1 hour on Day 11 | 4.4 (2.2) | 2.9 (0.9) | 4.9 (2.5) | 6.4 (1.7) | 9.7 (2.4) | NA (NA) — tests not performed
  Tumor Necrosis Factor ἁ - 2 hours on Day 11 | 1.9 (0.6) | 4 (3.8) | 4 (1.9) | 4.7 (3) | 9 (2.1) | NA (NA) — tests not performed
  Tumor Necrosis Factor ἁ - 4 hours on Day 11 | 2.7 (0.9) | 2.9 (1.3) | 5 (2.7) | 5.4 (1) | 7.7 (2) | NA (NA) — tests not performed
  Tumor Necrosis Factor ἁ - 12 hours on Day 11 | NA (NA) — tests not performed | NA (NA) — tests not performed | NA (NA) — tests not performed | NA (NA) — tests not performed | NA (NA) — tests not performed | NA (NA) — tests not performed
  Tumor Necrosis Factor ἁ - 24 hours on Day 12 | 2.3 (0.6) | 2.8 (1) | 15.4 (20) | 3.5 (0.7) | 5 (1.4) | NA (NA) — tests not performed

10. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 18 months (m)/27 days(d), 3 m, 9 m/13d, 15 m/20d, 28 m/17d, 1 m/23d, 15 m/8d, 4 m/5d, and 6 m/30d for levels 1-9 respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Level 1 - 0.1 mcg/kg/Day x 10 Days | Dose Escalation Level 2 - 0.25 mcg/kg/Day x 10 Days | Dose Escalation Level 3 - 0.5 mcg/kg/Day x 10 Days | Dose Escalation Level 4 - 1 mcg/kg/Day x 10 Days | Dose Escalation Level 5 - 2 mcg/kg/Day x 10 Days | Dose Escalation Level 6 - 4 mcg/kg/Day x 10 Days | Dose Escalation Level 7 - 3 mcg/kg/Day x 5 Days | Dose Escalation Level 8 - 4 mcg/kg/Day x 5 Days | Dose Escalation Level 9 - 5 mcg/kg/Day x 5 Days
Number analyzed (Participants) | 4 | 3 | 3 | 6 | 9 | 2 | 4 | 3 | 4
Participants | 4 | 3 | 3 | 6 | 9 | 2 | 4 | 3 | 4

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 18 months and 27 days for level 1, 3 months for level 2, 9 months and 13 days for level 3, 15 months and 20 days for level 4, 28 months and 17 days for level 5, 1 month and 23 days for level 6, 15 months and 8 days for level 7, 4 months and 5 days for level 8, and 6 months and 30 days for level 9.
Arm/Group | Dose Escalation Level 1 - 0.1 mcg/kg/Day x 10 Days | Dose Escalation Level 2 - 0.25 mcg/kg/Day x 10 Days | Dose Escalation Level 3 - 0.5 mcg/kg/Day x 10 Days | Dose Escalation Level 4 - 1 mcg/kg/Day x 10 Days | Dose Escalation Level 5 - 2 mcg/kg/Day x 10 Days | Dose Escalation Level 6 - 4 mcg/kg/Day x 10 Days | Dose Escalation Level 7 - 3 mcg/kg/Day x 5 Days | Dose Escalation Level 8 - 4 mcg/kg/Day x 5 Days | Dose Escalation Level 9 - 5 mcg/kg/Day x 5 Days
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/3 | 1/6 | 0/9 | 1/2 | 0/4 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/3 | 1/3 | 3/6 | 2/9 | 2/2 | 0/4 | 1/3 | 2/4
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 3/3 | 6/6 | 9/9 | 2/2 | 4/4 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Level 1 - 0.1 mcg/kg/Day x 10 Days (N=4) | Dose Escalation Level 2 - 0.25 mcg/kg/Day x 10 Days (N=3) | Dose Escalation Level 3 - 0.5 mcg/kg/Day x 10 Days (N=3) | Dose Escalation Level 4 - 1 mcg/kg/Day x 10 Days (N=6) | Dose Escalation Level 5 - 2 mcg/kg/Day x 10 Days (N=9) | Dose Escalation Level 6 - 4 mcg/kg/Day x 10 Days (N=2) | Dose Escalation Level 7 - 3 mcg/kg/Day x 5 Days (N=4) | Dose Escalation Level 8 - 4 mcg/kg/Day x 5 Days (N=3) | Dose Escalation Level 9 - 5 mcg/kg/Day x 5 Days (N=4)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Duodenal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Recurrent retropharyngeal infection/abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, Direct bilirubin (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, Cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papilledema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden death NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visceral arterial ischemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Level 1 - 0.1 mcg/kg/Day x 10 Days (N=4) | Dose Escalation Level 2 - 0.25 mcg/kg/Day x 10 Days (N=3) | Dose Escalation Level 3 - 0.5 mcg/kg/Day x 10 Days (N=3) | Dose Escalation Level 4 - 1 mcg/kg/Day x 10 Days (N=6) | Dose Escalation Level 5 - 2 mcg/kg/Day x 10 Days (N=9) | Dose Escalation Level 6 - 4 mcg/kg/Day x 10 Days (N=2) | Dose Escalation Level 7 - 3 mcg/kg/Day x 5 Days (N=4) | Dose Escalation Level 8 - 4 mcg/kg/Day x 5 Days (N=3) | Dose Escalation Level 9 - 5 mcg/kg/Day x 5 Days (N=4)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (2) | 0 (0) | 2 (2) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (2) | 2 (2) | 1 (2) | 5 (26) | 7 (12) | 2 (2) | 2 (5) | 3 (8) | 4 (7)
Alkaline phosphatase increased (Investigations) | 1 (2) | 2 (5) | 0 (0) | 3 (14) | 9 (17) | 2 (5) | 1 (6) | 3 (12) | 4 (6)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (10) | 2 (4) | 2 (13) | 6 (37) | 9 (56) | 1 (3) | 2 (14) | 3 (9) | 3 (7)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 1 (2) | 1 (2) | 5 (29) | 7 (16) | 2 (4) | 2 (9) | 3 (6) | 4 (8)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (7) | 2 (7) | 2 (6) | 2 (5) | 2 (6) | 2 (4)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (3) | 1 (1) | 1 (1) | 2 (4) | 5 (6) | 0 (0) | 2 (8) | 2 (3) | 3 (4)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 4 (11) | 2 (7) | 1 (2) | 0 (0) | 2 (8) | 4 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 1 (1) | 2 (3) | 1 (1) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 1 (1) | 1 (2) | 3 (5) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Fever (General disorders) | 2 (4) | 2 (6) | 1 (5) | 5 (12) | 8 (20) | 2 (2) | 4 (14) | 3 (6) | 4 (10)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Mouth sores (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Oral ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, angular cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, Apthous ulcer (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 1 (4) | 2 (3) | 3 (6) | 3 (3) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (4) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (4) | 2 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 1 (2) | 3 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (8) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (9) | 2 (5) | 2 (7) | 6 (59) | 9 (50) | 2 (5) | 2 (14) | 3 (18) | 4 (14)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 1 (1) | 4 (5) | 3 (5) | 0 (0) | 1 (1) | 1 (3) | 4 (5)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (7) | 3 (3) | 5 (9) | 1 (3) | 4 (6) | 1 (1) | 4 (10)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (4) | 1 (2) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 4 (5)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (5) | 4 (10) | 3 (15) | 1 (3) | 2 (2) | 3 (6) | 3 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (6) | 4 (10) | 2 (3) | 4 (7) | 3 (6) | 3 (10)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, Cold-like symptoms (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Investigations - Other, Direct bilirubin (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (18) | 3 (7) | 3 (23) | 6 (48) | 9 (46) | 2 (7) | 2 (17) | 3 (20) | 4 (17)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 6 (12) | 8 (14) | 1 (1) | 1 (3) | 3 (7) | 3 (6)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 7 (9) | 1 (1) | 2 (2) | 2 (4) | 3 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (5) | 2 (4) | 6 (21) | 0 (0) | 1 (2) | 2 (6) | 2 (2)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (3) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (4) | 2 (9) | 2 (5) | 3 (10) | 7 (16) | 2 (4) | 2 (8) | 3 (5) | 3 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (7) | 0 (0) | 2 (4) | 0 (0) | 2 (3)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Erythema, bilateral cheeks (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Facial erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Hands and Feet, Skin Sloughing (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Skin Peeling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, erythema to cheeks (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 1 (3) | 2 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (3) | 2 (5) | 3 (11) | 2 (3) | 6 (23) | 1 (1) | 2 (14) | 2 (16) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT01572493/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT01572493/ICF_001.pdf